CLINICAL TRIAL: NCT05357794
Title: Effectiveness of Concurrent Ultra-Low-Dose Total-Skin Electron Beam Therapy and Brentuximab Vedotin Given Quarterly Over 12 Months for Patients With Mycosis Fungoides
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0500; NCI-2022-03831 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brentuximab vedotin (Experimental): Participant will receive radiation therapy to the entire skin surface over the course of 2 days. Each dose will take about 60 to 90 minutes and will vary from one patient to another
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin — Given by Vein (IV)
  Other Names: SGN-35; Adcetris

SUMMARY:
To learn if a form of radiation therapy (called ultra-low-dose - total skin electron beam therapy [ULD-TSEBT]) in combination with brentuximab vedotin can help to control mycosis fungoides

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective:

The primary objective is to determine the overall response rate (ORR), to ultra-low-dose-total-skin electron beam therapy with brentuximab vedotin (ULD-TSEBT+BV) among patients with stage I-IV mycosis fungoides/Sezary syndrome.

Secondary Objective:

Key secondary objective is to determine the time to treatment failure (TTF) Determine the safety of brentuximab vedotin (BV) with fractionated ultra-low-dose-total-skin electron beam therapy (ULD-TSEBT) Describe the rate and grade of neuropathy associated with lower-dose BV by using CTCAE V5.0 Assess quality of life by using the validated Skindex-29 instrument and FACT instrument Determine the complete response rate (CRR) Determine progression-free survival (PFS) Determine overall survival (OS) Note: The study follow up timeframe for CRR, PFS and OS is expected to be two and half years.

Assess the relationship between ORR and CD30 expression level

Exploratory Objectives:

Objective: To identify tumor and peripheral blood markers that predict response to concurrent BV with fractionated ULD-TSEBT, including SS component in the history.

Objective: Identification of tumor and peripheral blood markers that are predictive of response to the combination therapy. Define changes in the TCR clonotypes, phenotypes, and inflammatory cytokine levels in biopsy specimens, peripheral blood leukocytes, and serum. Correlate changes in anti-tumor immune responses with clinic-pathological variables and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-confirmed mycosis fungoides in stage I-IV (APPENDICES 3 AND 4); the presence of Sezary cells in the blood is acceptable at original diagnosis or at enrollment into the protocol, as long as the patient has current mycosis fungoides in the skin and the sesary cells in peripheral blood are < 1000 cells/ microlitre at the time of enrollment.
2. Participants with relapsed/ refractory mycosis fungoides expressing at least 1% CD30 are eligible.
3. Previous systemic anticancer therapy must have been discontinued at least 1 week before treatment
4. In the case of myelosuppressive chemotherapy treatment may start once counts have recovered including absolute WBC> 1000, platelets> 50K.
5. Topical or systemic steroids (equivalent to 10 mg/day of prednisone) may be considered if the dose of such steroids has been constant and their discontinuation may lead to rebound flare in disease, adrenal insufficiency, and/or unnecessary suffering, after discussion with the Principal Investigator.
6. 18 years of age or older
7. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 3 (APPENDIX 5)
8. No required wash-out period for prior therapies
9. HIV+ participants must be on stable antiretroviral treatment for 12 weeks before the first day of cycle 1 (C1D1), with CD4 count >200 within the 7 days before C1D1.
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Concurrent use of other systemic anticancer agents or treatments (including steroids unless adrenal insufficiency has been diagnosed) for mycosis fungoides or Sezary syndrome
2. Grade 2 or greater neuropathy
3. Severe renal impairment (creatinine clearance [CrCL] <30 mL/min)
4. Moderate or severe hepatic impairment (Child-Pugh B or C; see APPENDIX 6 for ChildPugh classification chart)
5. Women of reproductive potential must have a negative serum ß human chorionic gonadotropin (ß-HCG) pregnancy test within 1 week of C1D1. They should discuss contraception with the treating provider. And agree to use adequate birth control measures (oral, implanted, or barrier methods) while on study Female participants of childbearing potential who are not abstinent and intend to be sexually active with a non sterilized male partner must use at least 1 highly effective method of contraception (Failure rate of <1% per year when used consistently and correctly) throughout the total duration of the drug treatment and the drug washout period as determined by your physician. Non-sterilized male partners of a female participants of childbearing potential must use male condom plus spermicide throughout this period. Cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Female participants should also refrain from breastfeeding throughout this period. Highly effective contraceptive methods:

   * Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation

     * oral
     * intravaginal
     * transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation

     * oral
     * injectable
   * Implantable progestogen-only hormonal contraception associated with inhibition of ovulation b
   * Intrauterine device (IUD)c
   * Intrauterine hormone-releasing system (IUS)c
   * Bilateral tubal occlusion
   * Surgical Sterilization
6. Receipt of systemic therapy for another primary malignancy (other than T-cell lymphoma). Participants with more than one type of lymphoma may be enrolled after discussion with the Principal Investigator
7. Underlying medical conditions including unstable cardiac disease, or other serious illness that would impair the ability of participants to undergo treatment
8. Any other medical history, including laboratory results, deemed by the Principal Investigator to be likely to interfere with participants participation in the study
9. Use of strong CYP3A4 inhibitors or inducers, or P-gp inhibitors, should be avoided given the potential effect on exposure to monomethyl auristatin E.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
To establish the overall response rate (ORR) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bouthaina Dabaja, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org